CLINICAL TRIAL: NCT01106937
Title: Risk Factors for Perioperative Pulmonary Embolism in Neurosurgical Patients in Respect of Factor XIII Activity
Brief Title: Factor XIII and Pulmonary Embolism in Neurosurgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Dr. Stefan Grau, Department of Neurosurgery, LMU Munich
Other Study IDs: SG-1
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-03

CONDITIONS: Brain Tumor; Vascular Lesion; Factor XIII Deficiency; Pulmonary Embolism
MeSH Terms: conditions — Brain Neoplasms; Factor XIII Deficiency; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with low Factor XIII: Postoperative occurence of pulmonary embolism in patients scheduled to undergo a neurosurgical procedure with laboratory-confirmed low levels of Factor XIII

SUMMARY:
Two studies (Gerlach et al. 2000; Gerlach et al. 2002) described the impact of factor XIII on the risk of prospective hemorrhage for patients undergoing craniotomy. Since then, factor XIII is measured and substituted in various centers. Few reports support the idea of factor XIII being involved in the formation of deep venous thrombosis and pulmonary embolism. In this prospective observational study, patients undergoing craniotomy for brain tumors or vascular lesions are investigated concerning the incidence of postoperative pulmonary embolism in respect of possible risk factors (factor XIII activity levels, standard coagulation parameters, tumor entity, blood loss).

ELIGIBILITY:
Inclusion Criteria:

* preoperatively low Factor XIII activity
* neurosurgical procedure (craniotomy)
* substitution of Factor XIII
* postoperative occurence of pulmonary embolism

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neurosurgical patients with a postoperative occurence of pulmonary embolism in with laboratory-confirmed preoperatively low levels of Factor XIII
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of pulmonary embolisms following Factor XIII substitution | 38 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Grau, Dr., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Department of Neurosurgery, LMU, Munich, Bavaria, Germany